CLINICAL TRIAL: NCT02714322
Title: Multicenter, Double-Blind, Randomized, 2-Arm, Parallel-Group, Equivalence Study Evaluating Efficacy and Safety Similarity of Mylan Adalimumab (MYL-1401A) Compared With Humira® in Subjects With Moderate-to-Severe Chronic Plaque Psoriasis
Brief Title: MYL-1401A Efficacy and Safety Comparability Study to Humira®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Mylan GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MYL-1401A-3001; 2014-003420-46 (EudraCT Number)
Record Dates: First submitted 2015-11-09; First posted 2016-03-21 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Psoriasis; Arthritis, Psoriatic
Keywords: Adalimumab; Biologics; Biosimilar
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MYL-1401A (Adalimumab) (Experimental): MYL-1401A initial dose of 80 mg administered subcutaneously (sc), followed by 40 mg sc given every other week starting 1 week after the initial dose
  Interventions: Biological: MYL-1401A (Adalimumab)
- Humira® (Adalimumab) (Active Comparator): Humira® initial dose of 80 mg administered subcutaneously (sc), followed by 40 mg sc given every other week starting 1 week after the initial dose
  Interventions: Biological: Humira® (Adalimumab)

INTERVENTIONS:
Biological: MYL-1401A (Adalimumab) — MYL-1401A initial dose of 80 mg administered subcutaneously (sc), followed by 40 mg sc given every other week starting 1 week after the initial dose
  Arms: MYL-1401A (Adalimumab)
Biological: Humira® (Adalimumab) — Humira® initial dose of 80 mg administered sc, followed by 40 mg sc given every other week starting 1 week after the initial dose
  Arms: Humira® (Adalimumab)

SUMMARY:
To assess the equivalence of MYL-1401A to Humira® with regards to efficacy in subjects with moderate-to-severe chronic plaque psoriasis

DETAILED DESCRIPTION:
Eligible subjects will be randomly assigned based on predefined stratification factors of weight, geographic region, and presence of psoriatic arthritis:

Randomization is 2:1 to MYL-1401A or Humira®, respectively.

The study will be conducted in the outpatient setting and comprises 3 periods: a screening period of up to 4 weeks, a 52-week treatment period, and a safety follow-up for 8 weeks.

A subject will be considered to have completed the study once they have completed the 52-week treatment period and the 8-week follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed the informed consent form
2. Subject is aged 18 to 75 years, inclusive, at time of Screening
3. Subject has had moderate-to-severe chronic plaque psoriasis for at least 6 months

   * Subject has involved BSA ≥10%, PASI ≥12, and sPGA ≥3 (moderate) at Screening and at Baseline
4. Subject has had stable disease for at least 2 months (i.e. without significant changes as defined by the investigator)
5. Subject is a candidate for systemic therapy
6. Subject has had a previous failure, inadequate response, intolerance, or contraindication to at least 1 conventional antipsoriatic systemic therapy
7. Subject is naïve to adalimumab therapy, approved or investigational
8. For females of childbearing potential, a negative serum pregnancy test during Screening and a negative urine pregnancy test at Baseline

Exclusion Criteria:

1. Subject diagnosed with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis, other skin conditions (e.g. eczema), or other systemic autoimmune disorder inflammatory disease at the time of the screening visit that would interfere with evaluations of the effect of the study treatment on psoriasis
2. Subject has used any of the following medications within specified time periods or will require their use during the study:

   * Topical medications within 2 weeks before the end of the screening period
   * oral psoralen with ultraviolet A (PUVA) phototherapy and/or ultraviolet B (UVB) phototherapy within 4 weeks before the end of the screening period
   * Nonbiologic systemic therapies within 4 weeks before the end of the screening period (e.g. cyclosporine, methotrexate, and acitretin)
   * Any prior or concomitant adalimumab therapy, approved or investigational
   * Any other investigational agent within 90 days or 5 half-lives of Screening (whichever is longer)
   * Any systemic steroid in the 4 weeks before the end of the screening period Note: Low-potency topical corticosteroids applied to the palms, soles, face, and intertriginous areas are permitted during study participation
3. Subject has received live vaccines during the 4 weeks prior to Screening or has the intention of receiving a live vaccine at any time during the study
4. Subject has a positive test for tuberculosis (TB) during Screening or a known history of active or latent TB, except documented and complete adequate treatment of TB or initiation (>1 month) of adequate prophylaxis of latent TB, with an isoniazid-based regimen

   * Subjects with a positive purified protein derivative (PPD) and a history of Bacillus Calmette-Guérin vaccination are allowed with a negative Interferon-γ release assays (IGRA)
   * Subjects with a positive PPD test without a history of Bacillus Calmette-Guérin vaccination or subjects with a positive or indeterminate IGRA are allowed if they have all of the following:
   * No symptoms or signs of active TB, including a negative chest x-ray within 3 months prior to the first dose of study treatment
   * Documented history of completion of adequate treatment of TB or initiation (>1 month) of adequate prophylaxis of latent TB, with an isoniazid-based regimen prior to receiving study treatment in accordance with local recommendations
5. Underlying condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious, or gastrointestinal) which, in the opinion of the investigator, significantly immunocompromises the subject and/or places the subject at unacceptable risk for receiving an immunomodulatory therapy
6. Subject has a planned surgical intervention during the duration of the study except those related to the underlying disease and which, in the opinion of the investigator, will not put the subject at further risk or hinder the subject's ability to maintain compliance with study treatment and the visit schedule
7. Subject has an active and serious infection or history of infections as follows:

   * Any active infection:
   * For which nonsystemic anti-infectives were used within 4 weeks prior to randomization.
   * Requiring hospitalization or systemic anti-infectives within 8 weeks prior to randomization
   * Recurrent or chronic infections or other active infection that, in the opinion of the investigator, might cause this study to be detrimental to the subject
   * Invasive fungal infection or mycobacterial infection
   * Opportunistic infections, such as listeriosis, legionellosis, or pneumocystis
8. Subject is positive for human immunodeficiency virus, hepatitis C virus antibody or hepatitis B surface antigen (HBsAg) or is positive for hepatitis B core antibody and negative for HBsAg at Screening
9. Subject has a history of clinically significant hematological abnormalities, including cytopenias (e.g. thrombocytopenia, leukopenia)
10. Subject has severe progressive or uncontrolled, clinically significant disease that in the judgment of the investigator renders the subject unsuitable for the study
11. Subject has history of malignancy within 5 years except adequately treated cutaneous squamous or basal cell carcinoma, in situ cervical cancer or in situ breast ductal carcinoma
12. Subject has active neurological disease such as multiple sclerosis, Guillain-Barré syndrome, optic neuritis, transverse myelitis, or history of neurologic symptoms suggestive of central nervous system demyelinating disease
13. Subject has moderate-to-severe heart failure (New York Heart Association class III/IV)
14. Subject has a history of hypersensitivity to the active substance or to any of the excipients of Humira® or MYL-1401A
15. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation
16. Evidence of alcohol or drug abuse or dependency at the time of Screening, for the 5 years prior to Screening or during the study
17. Subject is unable to follow study instructions and comply with the protocol in the opinion of the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Percent improvement in PASI from Baseline | Baseline and Week 12

SECONDARY OUTCOMES:
Proportion of subjects showing at least a 75% improvement in PASI (PASI 75 response rate) | Week 12
Number of subjects achieving static Physician's Global Assessment (sPGA) responses of clear (0) or almost clear (1) | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Abhijit Barve, MD, Study Chair — Mylan
Locations (33):
- Bulgaria (5):
  - Mylan Investigational Site 102, Plovdiv
  - Mylan Investigational Site 105, Plovdiv
  - Mylan Investigational Site 101, Sevlievo
  - Mylan Investigational Site 100, Sofia
  - Mylan Investigational Site 103, Sofia
- Estonia (6):
  - Mylan Investigational Site 107, Tallinn
  - Mylan Investigational Site 108, Tallinn
  - Mylan Investigational Site 109, Tallinn
  - Mylan Investigational site 110, Tallinn
  - Mylan Investigational Site 106, Tartu
  - Mylan Investigational SIte 112, Tartu
- Hungary (5):
  - Mylan Investigational Site 127, Budapest
  - Mylan Investigational Site 128, Budapest
  - Mylan Investigational Site 125, Debrecen
  - Mylan Investigational Site 129, Gyula
  - Mylan Investigational Site 126, Szekszárd
- Poland (11):
  - Mylan Investigational Site 131, Bialystok
  - Mylan Investigational Site 137, Bialystok
  - Mylan Investigational Site 135, Iwonicz-Zdrój
  - Mylan Investigational Site 140, Krakow
  - Mylan Investigational Site 139, Lodz
  - Mylan Investigational Site 133, Olsztyn
  - Mylan Investigational Site 138, Poznan
  - Mylan Investigational Site 136, Warsaw
  - Mylan Investigational Site 130, Wroclaw
  - Mylan Investigational Site 132, Wroclaw
  - Mylan Investigational Site 134, Wroclaw
- Russia (4):
  - Mylan investigational site 156, Kazan'
  - Mylan Investigational site 155, Penza
  - Mylan Investigational Site 148, Ryazan
  - Mylan Investigational Site 149, Saint Petersburg
- Ukraine (2):
  - Mylan Investigational site 159, Kharkiv
  - Mylan investigational site 161, Uzhhorod

IPD SHARING:
Plan to Share IPD: No